CLINICAL TRIAL: NCT01060982
Title: Observation of Histological Changes in Parathyroid Adenomas Following High Intensity Focused Ultrasound (HIFU)Treatment Procedure: A Monocentre, Open, Uncontrolled Study
Brief Title: Observation of Histological Changes in Parathyroid Adenomas Following High Intensity Focused Ultrasound (HIFU) Treatment Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theraclion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HIFU/F/12.02
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Primary Parathyroid Adenomas
Keywords: Primary hyperparathyroidism; High Intensity Focused Ultrasound; Parathyroid tumor; Parathyroid hormone; Calcium
MeSH Terms: conditions — Hyperparathyroidism, Primary; Parathyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HIFU treatment (Experimental)
  Interventions: Device: Ultrasonic ablation device

INTERVENTIONS:
Device: Ultrasonic ablation device — One High Intensity focused ultrasound session before surgery. Use of appropriate energy for each patient
  Other Names: TH-One

SUMMARY:
This study is a multicentre, open, uncontrolled trial for the observation of histological changes in parathyroid adenomas following high intensity focused ultrasound (HIFU).

This study will be conducted in France in 10 patients with primary hyperparathyroidism scheduled for a parathyroidectomy. The patient will receive an HIFU treatment in the center of the adenoma before the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient 18 years or older.
* Patients with diagnosed primary hyperparathyroidism (clinical symptoms and/or biochemical disturbances) scheduled for parathyroidectomy.
* One diseased parathyroid gland, visualized by ultrasonography.
* The diseased targeted parathyroid gland accessible for HIFU treatment (anonymised ultrasonographic images to be sent to the sponsor's technical team for validation).
* Normal pretreatment nasofibroscopy.
* Voluntary signed informed consent.

Exclusion Criteria:

* Inaccessibility or high risk of targeting neighbouring structures, as evidenced by:

  * Targeted area located less than 2 mm laterally from the oesophagus or the carotid artery
  * Targeted area located less than 3 mm laterally from the trachea,
  * Significant hyperechoic area with a posterior shadow located less than 10 mm behind the targeted area (behind to be understood as posterior to the targeted area in the direction of the HIFU beam)
* Investigator appreciation of any abnormal blood test that could contraindicate treatment with HIFU (bleeding abnormalities)
* Known spondylitis of the neck vertebrae
* Head and/or neck disease that prevents hyperextension of neck.
* Known history of parathyroid or other neoplasias in the neck region.
* History of neck irradiation
* Patients whose concurrent illnesses, disability, or geographical residence would hamper attendance at required study visit
* Pregnant or lactating woman.
* Female patient of childbearing age if not having a suitable contraception method.
* Patients who have received any investigational drug or device within the last 15 days and/or patients who are currently participating in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Histology of excised gland. | After surgery performed the same day as High intensity focused ultrasound treatment

CONTACTS AND LOCATIONS:
Overall Officials: Philippe BONNICHON, MD, Principal Investigator — Cochin Hospital, Paris, Fance
Locations (2):
- France (2):
  - Hôpital Privé des Peupliers, Paris
  - Cochin Hospital, Paris